CLINICAL TRIAL: NCT05161442
Title: Minimally Invasive Surgery in Crohn's Disease: Laparoscopic vs Robotic
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David W. Larson, Principal Investigator, Mayo Clinic
Other Study IDs: 21-002141
Record Dates: First submitted 2021-10-11; First posted 2021-12-17 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease; Surgery
Keywords: crohn disease; minimally invasive surgery; ileocolic resection; outcomes; complication; enhanced recovery after surgery
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational cohort study including patients with Crohn's Disease undergoing minimally invasive ileocolic resection.

DETAILED DESCRIPTION:
All consecutive patients with Crohn's disease (CD) who underwent minimally invasive ileocolic resection from 2014 at Mayo Clinic were retrospectively identified using a prospectively maintained institutional database.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease
* Ileocolic resection

Exclusion Criteria:

- N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective cohort of patients with Crohn underwent ileocolic resection.
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2014-01; Primary Completion 2021-12-31 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
conversion | 30-day after surgery
  intraoperative conversion to open (yes/no)
postoperative complications | 30-day after surgery
  30-day postoperative complications described as binary variable (yes/no) and type.
postoperative complications grade | 30-day after surgery
  30-day postoperative complications graded according Clavien-Dindo classification (I-V).
length of hospital stay | 30-day after surgery
  length of hospital stay (days)
hospital readmission | 30-day after surgery
  30-day hospital readmission (yes/no)

SECONDARY OUTCOMES:
Recurrence date | 5 years
  Endoscopic recurrence (date)
Recurrence grade | 5 years
  Endoscopic recurrence (Rutgeerts)
Recurrence clinical | 5 years
  Clinical recurrence (yes/no)
Gastrointestinal Quality of Life Index | 7 years
  quality of life measured according to Gastrointestinal Quality of Life Index (GIQLI)

CONTACTS AND LOCATIONS:
Overall Officials: David W Larson, MD,MBA, Principal Investigator — Mayo Clinic, Rochester, MN

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to third part, according to the condition indicated in the IRB.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials